CLINICAL TRIAL: NCT00787033
Title: A Phase 1, Open-Label, Dose Escalation Study To Evaluate Safety, Pharmacokinetics And Pharmacodynamics Of PF-04554878 In Patients With Advanced Non-Hematologic Malignancies
Brief Title: A Study Of PF-04554878 In Patients With Advanced Non-Hematologic Malignancies
Acronym: B0761001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Verastem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B0761001
Record Dates: First submitted 2008-11-05; First posted 2008-11-07 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2013-03

CONDITIONS: Cancer
Keywords: Focal Adhesion Kinase; Advanced Non-Hematologic Malignancies
MeSH Terms: conditions — Neoplasms | interventions — defactinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Dose escalation study with Expansion Cohorts at RP2D and Schedule
  Interventions: Drug: PF-04554878

INTERVENTIONS:
Drug: PF-04554878 — Oral pills at increasing dose twice daily, 21 day cycle, continuous treatment schedule until progression of disease, unacceptable toxicity, or patient request. Some patients will undergo serial biopsy and/or FDG-PET imaging

SUMMARY:
Phase 1 safety, pharmacokinetics, and pharmacodynamics trial of the focal adhesion kinase (FAK) inhibitor PF-04554878 in patients with advanced non-hematologic malignancies, including patients with malignancies appropriate for serial biopsy. Screening consists of medical history, physical examination ECOG performance status, blood draws, a pregnancy test for female patients of childbearing potential, a FDG-PET and tumor imaging. Treatment consists of PF-04554878 pills continued until progression of disease, unacceptable toxicity, or patient request. Evaluations for bioactivity are measured by serial FDG-PET and blood tests for biomarkers related to FAK and Pyk2 activities.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced non-hematologic malignancies.
* Adequate organ function, including bilirubin less than 1.5 x ULN, and ECOG (Eastern Cooperative Oncology Group) performance status of 0-2.

Exclusion Criteria:

* Clinically significant gastrointestinal abnormalities, requirement for systemic anticoagulants or potent CYP 2C8 inhibitors, and history of clinically significant cardiac or pulmonary disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-12; Primary Completion 2011-03 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose | 18 months
Overall safety profile of PF-04554878, including Dose-Limiting Toxicity (DLT) | 18 months

SECONDARY OUTCOMES:
Tumor metabolic response | 18 months
PF-04554878 pharmacokinetic (PK) parameters and Midazolam PK parameters | 18 months
FAK-related biomarkers in tumor biopsies and blood | 18 months
Molecular profiling (genomics data) based on the optional studies with whole blood and/or tumor samples | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (2):
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Nashville, Tennessee
- Pfizer Investigational Site, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Jones SF, Siu LL, Bendell JC, Cleary JM, Razak AR, Infante JR, Pandya SS, Bedard PL, Pierce KJ, Houk B, Roberts WG, Shreeve SM, Shapiro GI. A phase I study of VS-6063, a second-generation focal adhesion kinase inhibitor, in patients with advanced solid tumors. Invest New Drugs. 2015 Oct;33(5):1100-7. doi: 10.1007/s10637-015-0282-y. Epub 2015 Sep 4. PMID 26334219
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0761001&StudyName=A%20Study%20Of%20PF-04554878%20In%20Patients%20With%20Advanced%20Non-Hematologic%20Malignancies%0A